CLINICAL TRIAL: NCT03548636
Title: If THEY Build it, Will THEY Act? Novel Approaches to Increasing Physical Activity Among Breast Cancer Survivors
Brief Title: Project MOVE: Increasing Physical Activity Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Cristina Caperchione, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H14-02502
Record Dates: First submitted 2018-05-08; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Cancer Prevention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Feasibility Study (Experimental): Participant determined 6-month physical activity program
  Interventions: Behavioral: Single-Arm Feasibility Study

INTERVENTIONS:
Behavioral: Single-Arm Feasibility Study — Groups of 8 to 12 participants, consisting of >50% breast cancer survivors, were invited to apply for up to $2000 to enable access to equipment, resources, facilities, instruction and/or transportation to implement a physical activity intervention. Applicants were assessed by a Grant Review Panel. Successful applicants were informed that they would receive an additional $500 incentive if they increased their group's mean physical activity at six month follow-up (assessed via accelerometry).

SUMMARY:
The purpose of this research is to implement and evaluate the feasibility of Project MOVE, a program aimed to increase physical activity among breast cancer survivors through microgrants and financial incentives.

DETAILED DESCRIPTION:
Despite the physical and psychological health benefits associated with physical activity for breast cancer survivors, up to 70% of female breast survivors are not meeting minimum recommended physical activity guidelines. The purpose of this research was to develop, implement and assess the feasibility of Project MOVE, an innovative approach to increase physical activity among breast cancer survivors through the use of Action Grants, a combination of microgrants (small amounts of money awarded to groups of individuals to support a physical activity initiative) and financial incentives. Twelve groups of 8-12 adult women who are breast cancer survivors (N=132) were recruited for the study via face-to-face meetings with breast cancer-related stakeholders, local print and radio media, social media, and pamphlets and posters at community organisations and medical clinics. Each group submitted a microgrant application outlining their proposed physical activity initiative. Successful applicants were determined by a grant review panel and informed of a financial incentive upon meeting their physical activity goals. Primary (program feasibility) and secondary (physical activity, quality of life, motivation to exercise and social connection) outcome measures were evaluated using a mixed-methods approach including focus groups, self-reported questionnaires, semi-structured telephone interviews and objective physical activity measures. Measures were collected at baseline, post-intervention (6 months) and 12-month follow-up. Findings from this study were used to asses the implementation and feasibility of Project MOVE as a strategy for increasing physical activity among breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivors
* 18+ years old,
* Residing in the Okanagan region of British Columbia, Canada

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

PRIMARY OUTCOMES:
Program Feasibility (questionnaire) | Post-intervention (6 months)
  Program feasibility will be evaluated using mixed-methods, including a questionnaire, focus groups and semi-structured telephone interviews. A 5-point Likert-scale questionnaire with 1 being "strongly disagree" and 5 being "strongly agree" will be one method used to measure feasibility. Questions will focus on program satisfaction, program appropriateness and participant's perceived confidence to engage in physical activity and continue to engage in physical activity in the long term.
Program Feasibility (focus groups) | Post-intervention (6 months)
  Program feasibility will also be measured using focus groups. Focus groups with each of the Project MOVE groups (ranging 8 to 12 participants per group) will be conducted at the 6-month follow-up. All group members will be invited to participate. Questions will pertain to participants' experiences of Project MOVE specific to adoption, implementation, and maintenance. The focus groups will be audio recorded with a digital SonyTM recorder (ICD-PX333) and transcribed verbatim.
Program Feasibility (interviews) | 1-4 weeks post-intervention 6 month follow-up
  Program feasibility will also be measured using semi-structured interviews with each of the group leaders. Phone interviews will be scheduled within 1-4 weeks after the 6-month follow-up data collection period. Open ended questions will be utilized and will focus on the microgrant application process, challenges and enablers to leading a Project MOVE group, and the leader's perception of group member's experiences with Project MOVE. Phone interviews will be recorded using the digital SonyTM recorder (ICD-PX333) and transcribed verbatim.

SECONDARY OUTCOMES:
Physical Activity Behaviour (Objective) | Baseline, Post-intervention (6 months) and 12-month follow-up
  Measured using an Actigraph GT3X™ accelerometer, which is the 'gold standard' measure of physical activity in adults. The Actigraph GT3X™ accelerometer was worn by all participants during all waking hours over 7 consecutive days. The accelerometers were initialised to record steps, inclination and acceleration counts in triaxial mode, using 60s epochs. Established cut-off points were used to calculate daily minutes of moderate (2691-6166 counts/min) and vigorous (>6167counts/min) physical activity while controlling for the number of days the accelerometer was worn. Data are included in the analyses if there are no extreme counts (>20000) and if data are available for at least 600min wear time per day on 5 days. Participants with invalid data were asked to wear the activity monitor for a further 7 days.
Physical Activity Behaviour (Subjective) | Baseline, Post-intervention (6 months) and 12-month follow-up
  Measured by self-report using a modified version of the Godin Leisure-Time Exercise Questionnaire (GLTEQ). Participants were asked to indicate the frequency and type of intensity (i.e. light, moderate, vigorous) of their daily physical activity per week and the duration (min) of these sessions. All responses were converted to minutes and calculated in accordance with the metabolic equivalent (MET) minutes method. A cut-off point of ≥600 MET minutes was used to dichotomise participants as 'adequately active for health benefit' or 'inadequately active'.
Anthropometrics | Baseline, Post-intervention (6 months) and 12-month follow-up
  Measured height and weight to calculate body mass index (BMI).
Sedentary Behaviour (Objective) | Baseline, Post-intervention (6 months) and 12-month follow-up
  Measured using Actigraph GT3X™ accelerometer (using a 30s epoch). Sedentary time was determined as <100 counts/min, adjusted for non-wear time operationalised as at least 60 min of consecutive zeros.
Sedentary Behaviour (Subjective) | Baseline, Post-intervention (6 months) and 12-month follow-up
  Measured by self-report using the Marshall Sitting Questionnaire (MSQ). The MSQ assesses time spent sitting on weekdays and weekend days at work, travelling and at home. Data from the sitting time questionnaire was used to create an estimate of total weekday and weekend-day sitting times (min/day) by summing the time reported in each domain (higher total hours are indicative of more time spent sedentary).
Quality of Life | Baseline, Post-intervention (6 months) and 12-month follow-up
  Assessed using the SF 36 Medical Outcomes Study Survey (SF-36/RAND 36), a 36-item tool used to measure overall quality of life across eight domains, including physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue and general health perceptions. Pre-coded numeric values are assigned to each scale, and all items are then scored on a 0 to 100 range, with a high score representing a more favourable health state. Additionally, items in each of the eight domains are averaged together to create eight separate domain scores.
Motivation to Engage in Exercise | Baseline, Post-intervention (6 months) and 12-month follow-up
  Measured using the Behavioral Regulation in Exercise Questionnaire-version 3 (BREQ-3). The BREQ-3 measures external regulation (e.g. 'I exercise because other people say I should'), introjected regulation (e.g. 'I feel guilty when I don't exercise'), identified regulation (e.g. 'I value the benefits of exercise') and intrinsic regulation (e.g. 'I exercise because it's fun') of exercise behaviour. Participant responses were scored using an item aggregation approach, which involves summarising participant responses by averaging the items of each individual subscale into six unique scores.
Social Support | Baseline, Post-intervention (6 months) and 12-month follow-up
  Assessed using the 6-item 'Positive Relationship with Others' subscale of the Ryff Scales of Psychological Well-being (RSPW), which measures multiple facets of psychological well-being. The subscale presents statements regarding one's personal relationships with others. Participants were asked to rate statements on a scale of 1-6, with 1 indicating strong disagreement and 6 indicating strong agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Caperchione, PhD, Principal Investigator — The University of British Columbia Okanagan

IPD SHARING:
Plan to Share IPD: No
Only the principal investigators and UBC research team members will have access to the raw data. CO-I's external to UBC will not require access to raw participant data. Any data that are shared will be aggregate data and have all identifiers removed. All of these individuals have training in issues concerning privacy, confidentiality, and are aware of their responsibilities to maintain these.

REFERENCES:
- [Derived] Caperchione CM, Sabiston CM, Stolp S, Bottorff JL, Campbell KL, Eves ND, Ellard SL, Gotay C, Sharp P, Pullen T, Fitzpatrick KM. A preliminary trial examining a 'real world' approach for increasing physical activity among breast cancer survivors: findings from project MOVE. BMC Cancer. 2019 Mar 27;19(1):272. doi: 10.1186/s12885-019-5470-2. PMID 30917793